CLINICAL TRIAL: NCT06480890
Title: A 12-Week Single-Cohort Study, to Evaluate Real-World Effectiveness of a Triple Combination Beclometasone Diproprionate/Formoterol Fumarate/Glycopyrronium Bromide (BDP/FF/GB) in a Single Pressurised Metered Dose Inhaler (Trimbow® pMDI) in Subjects With COPD
Brief Title: Real-World Effectiveness of a Triple Combination BDP/FF/GB in a Single Pressurised Metered Dose Inhaler in COPD Patients (TRIPHY)
Acronym: TRIPHY
Status: Completed | Type: Observational
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLI-05993AA1-23; CTR20241876 (Registry Identifier: Center for Drug Evaluation (China))
Record Dates: First submitted 2024-06-12; First posted 2024-06-28 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Lung functions; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to evaluate Real-World Effectiveness of a Triple Combination Beclometasone Diproprionate/Formoterol Fumarate/Glycopyrronium Bromide (BDP/FF/GB) in a Single Pressurised Metered Dose Inhaler (Trimbow® pMDI) in Subjects with Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
This real-world study is a multi-centre, single-cohort, ambi-directional observational cohort study with both retrospective and prospective data collection, with the primary objective to assess the 12-week effectiveness of BDP/FF/GB for COPD subjects in China. The index date is the initiation date of BDP/FF/GB, and subjects may have initiated treatment with BDP/FF/GB up to 12 weeks before enrolment. Baseline period is the 12 weeks prior to index date. The end of study (EOS) for each subject will be the earliest of the following: approximately 12 weeks after BDP/FF/GB initiation (the Week 12 Visit), BDP/FF/GB discontinuation plus 2 weeks, or at early withdrawal (such as consent withdrawal, death, or lost to follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are willing and able to give their written consent to participate in the study
2. Aged ≥40 years at BDP/FF/GB initiation
3. Had documented diagnosis of COPD prior to BDP/FF/GB initiation
4. Baseline CAT total score ≥10 (at the time of BDP/FF/GB initiation OR within the 12 weeks prior to treatment initiation, if no CAT total score is available on BDP/FF/GB initiation date)
5. Subjects who have initiated treatment with BDP/FF/GB within 12 weeks prior to informed consent form (ICF) signature, or on date of ICF signature

Exclusion Criteria:

1. Subjects who had been admitted to hospital for a COPD exacerbation within the last 4 weeks prior to BDP/FF/GB initiation
2. Subjects who are not likely to come back 12-weeks after BDP/FF/GB initiation, per Investigator judgement
3. Participation in any clinical trial in the 4 weeks prior to BDP/FF/GB initiation
4. Subjects had used any other single inhaler triple therapy before or at BDP/FF/GB initiation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with COPD (≥40 years and CAT total score ≥10) in China, who have newly initiated BDP/FF/GB without previous use of single inhaler triple therapy, and without recent hospitalisation for a COPD exacerbation. Detailed inclusion and exclusion criteria are listed below. Any treatment decision must have been taken prior to and independently of the subject's inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Effectiveness Measure | After 12-weeks of treatment with BDP/FF/GB on disease status
  COPD Assessment Test total score

SECONDARY OUTCOMES:
Effectiveness Measure | After 12-weeks of treatment with BDP/FF/GB
  Number and percentage of responders (i.e. subjects with a change from baseline in CAT total score ≤ -2) or non-responders (i.e. subjects with a change from baseline in CAT total score > -2 or with CAT total score at Week 12 missing).
Effectiveness Measure | After 12-weeks of treatment with BDP/FF/GB
  Mean absolute change from baseline in specific lung function parameter values (i.e. FEV1, FEV1 % of predicted, PEF) after 12 weeks of treatment with BDP/FF/GB.
Effectiveness Measure | After 12-weeks of treatment with BDP/FF/GB
  Mean absolute change from baseline in specific laboratory parameter values (i.e. eosinophil count) after 12 weeks of treatment with BDP/FF/GB.
Safety Measure | After 12-weeks of treatment with BDP/FF/GB
  Overall summary of AEs will be presented the number of subjects and percentage of subjects with any AEs.
Safety Measure | After 12-weeks of treatment with BDP/FF/GB
  Overall summary of adverse drug reactions (ADRs) will be presented with the number of subjects and percentage of subjects with any ADRs.
Safety Measure | After 12-weeks of treatment with BDP/FF/GB
  The number and percentage of subjects with any special situations will be summarised.

OTHER OUTCOMES:
Treatment Adherence | After 12-weeks of treatment with BDP/FF/GB
  Treatment adherence, by Test of Adherence to Inhaler (TAI)

CONTACTS AND LOCATIONS:
Overall Officials: Jinping Zheng, MD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (19):
- China (19):
  - Site 156119 - Peking University People's Hospital, Beijing, Beijing Municipality
  - Site 156110 Beijing Jingmei Group Genetal Hospital, Beijing, Beijing Municipality
  - Site 156101 - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Site 156113 - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Site 156114 - The Second Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Site 156108 - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Site 156125 - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Site 156117 - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Site 156109 - Shandong Provincial Hospital, Jinan, Shandong
  - Site 156122 - Deyang People's Hospital, Deyang, Sichuan
  - Site 156102 - Mianyang Central Hospital, Mianyang, Sichuan
  - Site 156121 - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang Uygur
  - Site 156106 - Huzhou Central Hospital, Huzhou, Zhejiang
  - Site 156115 - Jinhua Central Hospital, Jinhua, Zhejiang
  - Site 156124 - Lishui People's Hospital, Lishui, Zhejiang
  - Site 156112 - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - Site 156103 - Shaoxing People's Hospital, Shaoxing, Zhejiang
  - Site 156105 - Taizhou Central Hospital, Taizhou, Zhejiang
  - Site 156123 - Wenling People's Hospital, Wenling, Zhejiang

IPD SHARING:
Plan to Share IPD: No